CLINICAL TRIAL: NCT06613685
Title: An Operationally Seamless Phase 2/3, Randomized, Active-Controlled Study Evaluating the Safety and Efficacy of an Oral Weekly Regimen of GS-1720 in Combination With GS-4182 Versus Biktarvy in Treatment-Naive People With HIV-1
Brief Title: Study of Oral Weekly GS-1720 and GS-4182 Compared With Biktarvy in People With HIV-1 Who Have Not Been Treated
Acronym: WONDERS2
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-695-7156; 2024-512505-66 (Other: European Medicines Agency)
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Phase 2 of the study has 2 periods: Randomized and Extension, which are both open label.
  Phase 3 of the study has 2 periods: Randomized Period which would be double-blind (at least Week 96), followed by an Extension Period which will be Open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 2: GS-1720 + GS-4182 (Treatment Group 1) (Experimental): Participants will receive a 1-day loading dose of GS-1720 (1300 mg) and GS-4182 (600 mg) on Day 1.Thereafter, participants will take weekly doses of single agent GS-1720 (650 mg) and GS-4182 (300 mg) coadministered for at least 48 weeks.
  Interventions: Drug: GS-1720; Drug: GS-4182
- Phase 2: B/F/TAF (Treatment Group 2) (Active Comparator): Participants will receive B/F/TAF (50/200/25 mg) daily for at least 48 weeks.
  Interventions: Drug: Bictegravir/emtricitabine/tenofovir alafenamide
- Phase 2 Extension Phase: GS-1720/GS-4182 Fixed-dose Combination (FDC) (Experimental): At the end of the randomized treatment, Phase 2 participants will be given the option to participate in the Extension Phase. Phase 2 Treatment Group 1 will switch to GS-1720/GS-4182 FDC (650/300 mg) weekly. Phase 2 Treatment Group 2 will receive a loading dose of GS-1720/GS-4182 FDC (1300 mg/600 mg) on Extension Phase Day 1, then GS-1720/GS-4182 FDC (650/300 mg) weekly. Participants who choose to enter the Extension Phase will receive GS-1720/GS-4182 FDC tablets until the product becomes available or until Gilead Sciences elects to discontinue the study, whichever occurs first.
  Interventions: Drug: GS-1720/GS-4182 FDC
- Phase 3: GS-1720/GS-4182 FDC + Placebo to Match (PTM) B/F/TAF (Treatment Group 1) (Experimental): Participants will receive a 1-day loading dose of GS-1720/GS-4182 FDC on Day 1. Thereafter, participants will receive GS-1720/GS-4182 FDC tablets weekly + PTM B/F/TAF once daily. Participants will receive treatment for at least 96 weeks.
  Interventions: Drug: GS-1720/GS-4182 FDC; Drug: Placebo to Match BVY
- Phase 3: B/F/TAF + PTM GS-1720/GS-4182 FDC (Treatment Group 2) (Active Comparator): Participants will receive oral B/F/TAF daily along with PTM GS-1720/GS-4182 FDC weekly for at least 96 weeks. Additionally, participants will receive a 1-day loading dose of PTM GS-1720/GS-4182 on Day 1.
  Interventions: Drug: Bictegravir/emtricitabine/tenofovir alafenamide; Drug: Placebo to Match GS1720/GS-4182 FDC
- Phase 3 Extension Phase: GS-1720/GS-4182 Fixed-dose Combination (FDC) (Experimental): After the end of blinded treatment, Phase 3 participants will be given the option to participate in the Extension Phase. Phase 3 Treatment Group 1 will continue to receive GS-1720/GS-4182 FDC weekly while PTM B/F/TAF will be discontinued. Phase 3 Treatment Group 2 will switch to receive GS-1720/GS-4182 FDC tablets weekly. Participants in Treatment Group 2 will also receive a 1-day loading dose of GS-1720/GS-4182 FDC on Extension Phase Day 1.
  Participants who choose to enter the Phase 3 Extension Phase will receive GS-1720/GS-4182 FDC tablets until the product becomes available or until Gilead Sciences elects to discontinue the study, whichever occurs first.
  Interventions: Drug: GS-1720/GS-4182 FDC

INTERVENTIONS:
Drug: GS-1720 — Tablets administered orally without regard to food
  Arms: Phase 2: GS-1720 + GS-4182 (Treatment Group 1)
Drug: GS-4182 — Tablets administered orally without regard to food
  Arms: Phase 2: GS-1720 + GS-4182 (Treatment Group 1)
Drug: Bictegravir/emtricitabine/tenofovir alafenamide — Tablets administered orally without regard to food
  Other Names: Biktarvy ®
  Arms: Phase 2: B/F/TAF (Treatment Group 2); Phase 3: B/F/TAF + PTM GS-1720/GS-4182 FDC (Treatment Group 2)
Drug: GS-1720/GS-4182 FDC — Tablets administered orally without regard to food
  Arms: Phase 2 Extension Phase: GS-1720/GS-4182 Fixed-dose Combination (FDC); Phase 3 Extension Phase: GS-1720/GS-4182 Fixed-dose Combination (FDC); Phase 3: GS-1720/GS-4182 FDC + Placebo to Match (PTM) B/F/TAF (Treatment Group 1)
Drug: Placebo to Match BVY — Tablets administered orally without regard to food
  Arms: Phase 3: GS-1720/GS-4182 FDC + Placebo to Match (PTM) B/F/TAF (Treatment Group 1)
Drug: Placebo to Match GS1720/GS-4182 FDC — Tablets administered orally without regard to food
  Arms: Phase 3: B/F/TAF + PTM GS-1720/GS-4182 FDC (Treatment Group 2)

SUMMARY:
The goal of this clinical study is to learn more about the experimental drugs GS-1720 (an oral, long-acting integrase strand transfer inhibitor (INSTI)) and GS-4182 (a prodrug of Lenacapavir (LEN)); to compare the combination of GS-1720 and GS-4182 with the current standard-of-care treatment bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (Biktarvy), to see if the combination of GS-1720 and GS-4182 is safe and if it works for treating human immunodeficiency virus type 1 (HIV-1) infection in treatment-naive people with HIV-1 (PWH).

This study has two phases: Phase 2 and Phase 3.

The primary objectives of this study are:

Phase 2: To evaluate the efficacy of oral weekly GS-1720 coadministered with GS-4182 versus continuing Biktarvy (BVY) in treatment-naive PWH at Week 24.

Phase 3: To evaluate the efficacy of oral weekly GS-1720/GS-4182 fixed-dose combination (FDC) tablet regimen versus continuing BVY in treatment-naive PWH at Week 48.

ELIGIBILITY:
Key Inclusion Criteria:

* HIV-1 RNA ≥ 500 copies/mL at screening.
* Antiretroviral (ARV) treatment-naive, except the use of oral pre-exposure prophylaxis (PrEP) or postexposure prophylaxis (PEP) with emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) or F/TAF, up to 1 month prior to screening.

Key Exclusion Criteria:

* Prior use of any long acting parenteral antiretrovirals (ARVs) such as monoclonal antibodies, broadly neutralizing antibodies targeting HIV-1, LEN, injectable cabotegravir (including oral cabotegravir lead-in), and/or injectable rilpivirine.
* Documented resistance to the integrase strand-transfer inhibitor class, specifically, resistance-associated mutations E92G/Q, G118R, F121Y, Y143C/H/R, S147G, Q148H/K/R, N155H/S, or R263K in the integrase gene.
* Any of the following laboratory values at screening:

  1. CD4 cell count < 200 cells/mm3 at screening.
  2. Estimated glomerular filtrations arate < 60 mL/min according to the Modification of Diet in Renal Disease formula.
  3. Hepatic transaminases (aspartate aminotransferase and alanine aminotransferase) > 1.5 × upper limit of normal (ULN).
  4. Direct bilirubin > 1.5 × ULN.
  5. Platelets count < 50,000 cells/mm3.
  6. Hemoglobin < 8.0 g/dL.
* Active or occult hepatitis B virus infection.
* Active hepatitis C virus infection.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Proportion of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 as Determined by the United States (US) Food and Drug Administration (FDA)-defined Snapshot Algorithm | Week 24
Phase 3: Proportion of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm | Week 48

SECONDARY OUTCOMES:
Phase 2: Proportion of Participants With HIV-1 RNA < 50 copies/mL at Week 12 as Determined by the US FDA-defined Snapshot Algorithm | Week 12
Phase 2: Proportion of Participants With HIV-1 RNA < 50 copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm | Week 48
Phase 2: Change From Baseline in log10 HIV-1 RNA at Week 12 | Baseline, Week 12
Phase 2: Change From Baseline in log10 HIV-1 RNA at Week 24 | Baseline, Week 24
Phase 2: Change From Baseline in log10 HIV-1 RNA at Week 48 | Baseline, Week 48
Phase 2: Change From Baseline in Clusters of Differentiation 4 (CD4) Cell Count at Week 12 | Baseline, Week 12
Phase 2: Change From Baseline in CD4 Cell Count at Week 24 | Baseline, Week 24
Phase 2: Change From Baseline in CD4 Cell Count at Week 48 | Baseline, Week 48
Phase 2: Percentage of Participants Experiencing Treatment Emergent Adverse Events (TEAEs) Through Week 12 | First dose date up to Week 12
Phase 2: Percentage of Participants Experiencing TEAEs Through Week 24 | First dose date up to Week 24
Phase 2: Percentage of Participants Experiencing TEAEs Through Week 48 | First dose date up to Week 48
Phase 2: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities Through Week 12 | First dose date up to Week 12
Phase 2: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities Through Week 24 | First dose date up to Week 24
Phase 2: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities Through Week 48 | First dose date up to Week 48
Phase 2: Pharmacokinetic (PK) Parameter: Cmax of GS-1720 and Lenacapavir (LEN), as Applicable | Day 1 up to Week 24
  Cmax is defined as the maximum observed concentration of drug.
Phase 2: PK Parameter: Tmax of GS-1720 and LEN, as Applicable | Day 1 up to Week 24
  Tmax is defined as the time (observed time point) of Cmax.
Phase 2: PK Parameter: Ctau of GS-1720 and LEN, as Applicable | Day 1 up to Week 24
  Ctau is defined as the observed drug concentration at the end of the dosing interval.
Phase 2: PK Parameter: AUCtau of GS-1720 and LEN, as Applicable | Day 1 up to Week 24
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Phase 3: Proportion of Participants With HIV-1 RNA < 50 copies/mL at Week 96 as Determined by the US FDA-defined Snapshot Algorithm | Week 96
Phase 3: Change From Baseline in log10 HIV-1 RNA at Week 48 | Baseline, Week 48
Phase 3: Change From Baseline in log10 HIV-1 RNA at Week 96 | Baseline, Week 96
Phase 3: Change From Baseline in CD4 Cell Count at Week 48 | Baseline, Week 48
Phase 3: Change From Baseline in CD4 Cell Count at Week 96 | Baseline, Week 96
Phase 3: Percentage of Participants Experiencing TEAEs Through Week 48 | First dose date up to Week 48
Phase 3: Percentage of Participants Experiencing TEAEs Through Week 96 | First dose date up to Week 96
Phase 3: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities Through Week 48 | First dose date up to Week 48
Phase 3: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities Through Week 96 | First dose date up to Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (58):
- United States (21):
  - UAB 1917 Research Clinic, Birmingham, Alabama
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Mills Clinical Research, West Hollywood, California
  - Georgetown University Medical School, Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Emory University Hospital Midtown Infectious Disease Clinic, Atlanta, Georgia
  - Mercer University, Department of Internal Medicine, Macon, Georgia
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Michael's Medical Center, Newark, New Jersey
  - NYU Langone Health Vaccine Center, New York, New York
  - Medical University of South Carolina (MUSC) Research Nexus, Charleston, South Carolina
  - St Hope Foundation, Inc., Bellaire, Texas
  - Prism Health North Texas, Aids Arms, Dallas, Texas
  - North Texas Infectious Diseases Consultants, PA, Dallas, Texas
  - Texas Centers for Infectious Disease Associates, Fort Worth, Texas
  - UT Health San Antonio, San Antonio, Texas
  - MultiCare Rockwood Main Clinic, Spokane, Washington
- Canada (3):
  - Clinique Médicale L'Actuel, Montreal
  - Chronic Viral Illness Service / McGill University Health Centre, Montreal
  - Ottawa Hospital Research Institute, Ottawa
- Germany (5):
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik I, Immunologische Studienambulanz, Bonn
  - Universitätsmedizin Essen, Universitätsklinikum Essen, Klinik für Dermatologie, Venerologie und Allergologie, HPSTD-Ambulanz, Essen
  - ICH Study Center GmbH & Co. KG, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Rheumatologie und Immunologie, Gebäude K14, Hanover
  - Klinikum rechts der Isar, Technische Universität München, Klinik und Poliklinik für Innere Medizin II, München
- Poland (3):
  - Wojewódzki Szpital Obserwacyjno-Zakaźny im. Tadeusza Browicza, Bydoszcz
  - Punkt Zdrowia, Gdansk
  - Samodzielny Publiczny Wojewódzki Szpital Zespolony w Szczecinie, Szczecin
- Portugal (5):
  - Unidade Local de Saude de Amadora Sinatra EPE, Hospital Prof. Doutor Fernando Fonseca, Amadora
  - Unidade Local de Saúde de Lisboa Ocidental E.P.E. - Hospital Egas Moniz, Lisbon
  - Unidade Local de Saúde de Santo Maria E.P.E. - Hospital Santa Maria, Lisbon
  - Unidade Local de Saúde de Santo António, E.P.E., Porto
  - Unidade Local de Saúde de São João E.P.E., Porto
- Puerto Rico (2):
  - HOPE Clinical Research, San Juan, PR
  - Proyecto ACTU, San Juan, PR
- Romania (5):
  - Institutul National De Boli Infectioase Prof. Dr. Matei Bals, Bucharest
  - Spitalul Clinic De Urgenta Prof Dr Agrippa Ionescu, Bucharest
  - Spitalul Clinic De Boli Infectioase Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic de Boli Infectioase Constanta, Constanța
  - Clinical Hospital of Infectious Diseases and Pneumophysiology Dr. Victor Babes Timisoara, Timișoara
- South Africa (8):
  - JOSHA Research, Bloemfontein
  - Durban International Clinical Research Site, Enhancing Care Foundation, Durban
  - Synergy Biomed Research Institute, East London
  - CRISMO Research Center, Germiston
  - WITS RHI Research Centre, Johannesburg
  - Clinical Research Institute of South Africa (CRISA), KwaZulu-Natal
  - FPD Ndevana Community Research Site, Ndevana
  - The Aurum Institute Tembisa Clinic 4, Tembisa
- Spain (6):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Alvaro Cunqueiro, Pontevedra
  - Hospital Arnau de Vilanova de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06613685